CLINICAL TRIAL: NCT00411671
Title: A Phase II Study of Sorafenib (BAY 43-9006) in Chemorefractory Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: BATTLE Program: Sorafenib in Patients With NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0827
Record Dates: First submitted 2006-12-12; First posted 2006-12-14 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-01

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Non-Small Cell Lung Cancer; NSCLC; Sorafenib; BAY 43-9006; Battle Program
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib (Experimental): Sorafenib 400 mg By Mouth Twice Daily for 28 Days.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — 400 mg By Mouth Twice Daily for 28 Days.
  Other Names: BAY 43-9006

SUMMARY:
Primary Objective:

* To determine the 8 week progression-free survival rate (i.e. disease control rate) in patients with advanced non-small cell lung cancer (NSCLC) who have failed at least one prior chemotherapy regimen.

Secondary Objective:

The secondary objectives of this study will be to:

* Determine the overall response rate
* Determine the overall survival
* Determine the time to disease progression
* Assess the safety/toxicity of the study treatment
* Assess biomarker modulation in the tumor tissue and serum samples from the treatment.
* Assess plasma and intra-tumor concentrations of study treatment

DETAILED DESCRIPTION:
BAY 43-9006® (Sorafenib) is an experimental agent designed to stop the growth of cancer cells.

In order to enroll in this study, you must also be enrolled in Protocol 2005-0823: A Biomarker-integrated study in Chemorefractory patients with advanced Non-Small Cell Lung Cancer. Protocol 2005-0823 is the screening study in a group of studies called the BATTLE program. Participants in Protocol 2005-0823 are assigned to one of the treatment studies. The results of your tumor analysis helped the study doctor determine to assign you to this particular treatment study.

While on study, you will take 2 tablets of sorafenib each morning, and again each evening. Sorafenib should be taken with about 1 cup of water on an empty stomach (either 1 hour before a meal or 2 hours after a meal). Sorafenib must be swallowed whole without chewing. If you feel nauseated before or after taking the medication, anti-nausea medications should be used. If you miss a dose, you should skip it and take the next scheduled dose at the right time. Your medication should be stored at room temperature.

Every 4 weeks (1 cycle) your complete medical history will be recorded and you will have a physical exam, including measurement of vital signs (blood pressure, pulse, temperature, and breathing rate) and weight. Blood (about 2 teaspoons) and urine will be drawn for routine tests. You will have a performance status evaluation (questions about your ability to perform everyday activities) and blood drawn (about 1-2 teaspoons) to check your blood clotting function. Your study doctor will also ask you about any medications you are taking and your smoking history. You will be asked to record your weekly blood pressure for the first 6 weeks of study treatment. The study doctor or research nurse will review the log at each clinic visit.

Every 2 cycles, your tumor will be evaluated by chest x-ray and computed tomography (CT) or magnetic resonance imaging (MRI) scans to evaluate the status of the disease. If you are taking Coumadin® (warfarin), you will have blood drawn (about 1-2 teaspoons) to check your blood clotting function weekly for the first 6 weeks of treatment and then every cycle after that.

You may continue receiving sorafenib for as long as the cancer responds to study treatment. Your doctor may decide to take you off this study if you experience intolerable side effects or your medical condition gets worse. If you stop study treatment, you will be allowed to enroll in one of the remaining 3 protocols of the BATTLE program.

After you have stopped taking the study treatment, you will have a physical exam, including measurement of vital signs. Blood (about 2 teaspoons) and urine will be collected for routine tests. You will also have blood drawn (about 1-2 teaspoons) to check your blood clotting function. You will have a performance status evaluation, a chest x-ray, and a CT or MRI scan. Following this evaluation, you will be contacted by telephone every 3 months for up to 3 years, to see how you are doing.

You have the right to leave the study at any time. If you choose to stop participating in this study, you should contact the study chair and/or research nurse. Your doctor may decide to take you off this study if your medical condition gets worse and/or you are unable to comply with study requirements.

This is an investigational study. Sorafenib (BAY 43-9006) has been approved by the FDA for treatment of advanced renal cell cancer; however, it's use in this research study is investigational. Up to 62 patients will take part in this multicenter study. Up to 50 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a diagnosis of pathologically confirmed NSCLC by tumor biopsy and/or fine-needle aspiration.
2. The patient has a diagnosis of either stage IIIB, stage IV, or advanced, incurable NSCLC, and failed at least one front-line metastatic NSCLC chemotherapy regimen. (Patients who have failed adjuvant or locally advanced therapy within 6 months are also eligible to participate in study).
3. The patient has uni-dimensionally measurable NSCLC.
4. Karnofsky performance status >/= 60 or ECOG performance status 0-2
5. The patient has biopsy accessible tumor.
6. The patient has adequate hematologic function as defined by an absolute neutrophil count (ANC) >/= 1,500/mm^3, platelet count >/= 100,000/mm^3, white blood count (WBC) >/= 3,000/ mm^3, and hemoglobin >/= 9 g/dL.
7. The patient has adequate hepatic function as defined by a total bilirubin level </= 1.5 * the upper limit of normal, and alkaline phosphatase, AST or ALT </= 2.5 * the upper limit of normal.
8. The patient has adequate renal function as defined by a serum creatinine level </= 1.5 mg/dL or a calculated creatinine clearance of >/= 60cc/minute.
9. The patient has Prothrombin time (PT) < 1.5 * upper limit of normal
10. If patient has brain metastasis, they must have been stable (treated or asymptomatic) for at least 4 weeks after radiation if treated with radiation and not have used steroids for at least 1 week. Re-imaging performed after 2 weeks, upon completion of radiation therapy.
11. The patient is >/= 18 years of age.
12. The patient has signed informed consent.
13. The patient is eligible if disease free from a previously treated malignancy, other than a previous NSCLC, for greater than two years. Patients with a history of prior basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix are exempt from exclusion.
14. Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.Childbearing potential will be defined as women who have had menses within the past 12 months,who have not had tubal ligation or bilateral oophorectomy.Should a woman become pregnant or suspect that she is pregnant while participating in this study,she should inform her treating physician immediately.The patient,if a man,agrees to use effective contraception or abstinence.
15. Subject must be considered legally capable of providing his or her own consent for participation in this study.

Exclusion Criteria:

1. The patient has received prior investigational therapy, chemotherapy, surgery, or radiotherapy within 4 weeks of initiating study drug
2. The patient has undergone prior thoracic or abdominal surgery within 28 days of study entry, excluding prior diagnostic biopsy.
3. The patient has received radiation therapy to the measurable tumor within 6 months. Patients are allowed to have local irradiation for the management of tumor-related symptoms (bones, brain). However, if a patient has active new disease growing in the previously irradiated site, the patient will be eligible to participate in the study.
4. The patient has a significant medical history or unstable medical condition (unstable systemic disease: congestive heart failure (New York Heart Association Functional Classification class II or worse), recent myocardial infarction within 3 months, unstable angina, active infection (i.e. currently treated with antibiotics), uncontrolled hypertension). Patients with controlled diabetes will be allowed. Patient must be able to undergo procedure for tissue acquisition.
5. The patient has uncontrolled seizure disorder, active neurologic disease, or neuropathy >/= grade 2. Patients with meningeal or central nervous System (CNS) involvement by tumor are eligible for the study if the above exclusion criteria are not met.
6. The patient is pregnant (confirmed by serum b-HCG if applicable) or is breastfeeding.
7. Any condition that is unstable or could jeopardize the safety of the patient and its compliance in the study, in the investigator's judgment.
8. The patient is actively taking herbal remedies or over-the-counter biologics (e.g., shark cartilage, high dose antioxidants).
9. Patients will be allowed to have prior biologic (i.e. Vascular endothelial growth factor (VEGF), epidermal growth factor family (EGFR), etc.) therapy. However, the patient will be excluded from a given study if he/she has received the same therapy as the clinical trial (i.e. If a patient has been previously treated with bevacizumab, they are allowed to enroll in any of the 4 studies. If a patient has been previously treated with erlotinib, they are excluded from the clinical trials with erlotinib). In addition, if a patient has been previously treated with gefitinib (Iressa), they are excluded from the clinical trials with erlotinib.
10. Prior hemoptysis or bleeding diathesis.
11. Hypertension not controlled by medical therapy (systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg)
12. Known history of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C.
13. History of seizure disorder requiring medication (such as steroids or anti-epileptics).
14. History of organ allograft and bone marrow transplant
15. Previous malignancy (except for cervical carcinoma in situ, adequately treated basal cell carcinoma, or superficial bladder tumors [Ta, Tis & T1] or other malignancies curatively treated > 3 years prior to entry).
16. Patients with clinically significant bleeding (e.g., gastrointestinal bleeding) within the past month prior to study entry are ineligible.
17. Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 48 hours of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures (e.g., cervical cap, condom, and diaphragm) during the course of the trial. Oral birth control methods alone will not be considered adequate on this study, because of the potential pharmacokinetic interaction between BAY 43-9006 and oral contraceptives.
18. Substance abuse, medical, psychological or social conditions that, in the judgment of the investigator, is likely to interfere with the patient's participation in the study or evaluation of the study results.
19. Known allergy to the investigational agent or any agent given in association with this trial.
20. Concurrent use of St. John's Wort, Rifampicin, and/or ritonavir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2006-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Blumenschein, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Tam AL, Kim ES, Lee JJ, Ensor JE, Hicks ME, Tang X, Blumenschein GR, Alden CM, Erasmus JJ, Tsao A, Lippman SM, Hong WK, Wistuba II, Gupta S. Feasibility of image-guided transthoracic core-needle biopsy in the BATTLE lung trial. J Thorac Oncol. 2013 Apr;8(4):436-42. doi: 10.1097/JTO.0b013e318287c91e. PMID 23442309
- [Derived] Kim ES, Herbst RS, Wistuba II, Lee JJ, Blumenschein GR Jr, Tsao A, Stewart DJ, Hicks ME, Erasmus J Jr, Gupta S, Alden CM, Liu S, Tang X, Khuri FR, Tran HT, Johnson BE, Heymach JV, Mao L, Fossella F, Kies MS, Papadimitrakopoulou V, Davis SE, Lippman SM, Hong WK. The BATTLE trial: personalizing therapy for lung cancer. Cancer Discov. 2011 Jun;1(1):44-53. doi: 10.1158/2159-8274.CD-10-0010. Epub 2011 Jun 1. PMID 22586319
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: November 2006 to February 2010. All participants recruited at The University of Texas MD Anderson Cancer Center.
Groups:
- Sorafenib 400 mg: Sorafenib 400 mg by mouth twice daily in continuous 28 day cycles.
Period: Overall Study
Arm/Group | Sorafenib 400 mg
Started | 105
Completed | 85
Not Completed | 20
Not completed — Adverse Event | 15
Not completed — Death | 2
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib 400 mg
Number analyzed (Participants) | 105
Age, Customized [Number; unit: participants]
  < 60 years | 43
  >= 60 years | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 54
Region of Enrollment [Number; unit: participants]
  United States | 105

OUTCOME MEASURES:

1. Primary Outcome: 8-Week Disease Control Rate
Description: The disease control rate (DCR) was defined as the proportion of patients who did not meet Response Evaluation Criteria in Solid Tumors (RECIST) criteria for progressive disease (PD) at 8 weeks. Progressive disease was defined as at least a 20% increase in the sum of longest diameter (LD) of measured lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Baseline to 8 weeks
Population: Of the enrolled participants, 98 were evaluable for the outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Sorafenib 400 mg
Number analyzed (Participants) | 98
percentage of participants | 58.2

2. Secondary Outcome: Progression-Free Survival
Description: The Progression-Free Survival (PFS) was measured from date of randomization until progressive disease (PD) or death respectively.
Time Frame: From date of randomization until PD or death respectively, up to 3 years
Population: Of the enrolled participants, only 98 were evaluable for the outcome.
Measure: Median (Full Range); unit: months
Arm/Group | Sorafenib 400 mg
Number analyzed (Participants) | 98
months | 2.83 [1.87 to 3.55]

3. Secondary Outcome: Tumor Response Measured Every 8-weeks
Description: Tumor responses was measured according to RECIST criteria. Tumor responses were defined as: Partial Response (PR): at least a 30% decrease in the sum of longest diameter (LD) of target lesions taking as reference the baseline sum LD. Stable Disease (SD): steady state of disease. Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Progressive Disease (PD): at least a 20% increase in the sum of LD of measured lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: At baseline and then every 8 weeks until treatment discontinuation.
Population: Of the enrolled participants, only 98 were evaluable for the outcome.
Measure: Number; unit: participants
Arm/Group | Sorafenib 400 mg
Number analyzed (Participants) | 98
participants
  Patial Response | 0
  Stable Disease | 57
  Progressive Disease | 36
  Early Progression | 5

ADVERSE EVENTS:
Time Frame: Adverse events will be recorded for all patients from the time of consent until 30 days following the last dose of study treatment.
Description: Collection period: December 18, 2006 to November 13, 2010.
Arm/Group | Sorafenib 400 mg
Serious Adverse Events (participants affected / at risk) | 105/105
Other Adverse Events (participants affected / at risk) | 53/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib 400 mg (N=105)
Cerebrovascular ischemia (Nervous system disorders) | 5 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Death (General disorders) | 16 (16)
Ruptured Graft (General disorders) | 1 (1)
Perforated Gastric Ulcer (Gastrointestinal disorders) | 1 (1)
Mental Status Changed (Psychiatric disorders) | 1 (1)
Acute Deterioration of General Health (General disorders) | 1 (1)
Cardiac Troponin (Cardiac disorders) | 2 (2)
Itchy Reddened Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Mild Swelling of the Finger Joints (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder Perforation (Renal and urinary disorders) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 2 (2)
Pain, Breast Area (General disorders) | 1 (1)
Scrotal Abscess (Reproductive system and breast disorders) | 1 (1)
Hypotonic (Blood and lymphatic system disorders) | 1 (1)
Hypovolemic (Blood and lymphatic system disorders) | 1 (1)
Paroxysmal Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Non Functioning Right Kidney (Renal and urinary disorders) | 1 (1)
Perinephric Abscess (Renal and urinary disorders) | 1 (1)
Generalized Oedema (Blood and lymphatic system disorders) | 1 (1)
Decompensation Hydroelectrolytic (Blood and lymphatic system disorders) | 1 (1)
Confusion (Nervous system disorders) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Tenesmus (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Anal Pain (Gastrointestinal disorders) | 1 (1)
Inflammed Caecum (Gastrointestinal disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 8 (8)
Bartholin Cyst (Reproductive system and breast disorders) | 1 (1)
Abdominal Abscess (Gastrointestinal disorders) | 2 (2)
Gastrointestinal Perforation (Gastrointestinal disorders) | 1 (1)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Groin Abscess (Infections and infestations) | 1 (1)
Herpes Zoster (Infections and infestations) | 2 (2)
Hand Foot Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Ejection Fraction (Cardiac disorders) | 1 (1)
Septic Shock (Immune system disorders) | 3 (3)
Fatal Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 2 (2)
Fatal Disseminated Intravasular Coagulation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Melasma (Skin and subcutaneous tissue disorders) | 1 (1)
Partial Thromboplastin Time Increased (Blood and lymphatic system disorders) | 1 (1)
Bruising of Left Extremity (Skin and subcutaneous tissue disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Tetany (Musculoskeletal and connective tissue disorders) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
General Physical Health Deterioration (General disorders) | 3 (3)
Proximal Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Toxicoderma (Skin and subcutaneous tissue disorders) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1)
Epigastralgia (Gastrointestinal disorders) | 1 (1)
Carcinomatous Peritonitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Liver Carcinoma Ruptured (Hepatobiliary disorders) | 1 (1)
Hemianopsia (Eye disorders) | 1 (1)
ADH Secretion Abnormality (Endocrine disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Agitation (Nervous system disorders) | 1 (1)
Cadiogenic Shock (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1)
Chest Pain (General disorders) | 2 (2)
Acute Myeloid Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 2 (2)
Interstitial Infiltrates (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatal Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 2 (2)
Fatal Pustulosis (Skin and subcutaneous tissue disorders) | 1 (1)
Oversedation from Oxycontin (Nervous system disorders) | 1 (1)
Pseudomonas Stutzeri Sepsis (Infections and infestations) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Klebsiella Sepsis (Infections and infestations) | 2 (2)
Sepsis (Immune system disorders) | 6 (6)
Failure to Thrive (General disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Left Hemiparesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Loss of Consciousness (Nervous system disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Rupture of Hepatocellular Carcinoma (Hepatobiliary disorders) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2)
Cognitive Disturbance (Nervous system disorders) | 1 (1)
General Health Degradation (General disorders) | 5 (5)
Drowsiness (General disorders) | 1 (1)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 4 (4)
Volume Depletion (Metabolism and nutrition disorders) | 1 (1)
Acute Renal Insufficiency (Renal and urinary disorders) | 1 (1)
Colon Perforation (Gastrointestinal disorders) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Acute Pancreatitis (Endocrine disorders) | 1 (1)
Fatal Cardiopulmonary Decompensation (Cardiac disorders) | 1 (1)
Paralytic Ileus (Nervous system disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Streptococcus Positive (Infections and infestations) | 1 (1)
Transient Troponin I elevated (Cardiac disorders) | 1 (1)
Perianal Abscess (Gastrointestinal disorders) | 1 (1)
Hepatic Function Disorder (Hepatobiliary disorders) | 4 (4)
Vasculitis (Vascular disorders) | 1 (1)
LDH Increased (Metabolism and nutrition disorders) | 1 (1)
GGTP Increased (Hepatobiliary disorders) | 1 (1)
Cheilitis (Skin and subcutaneous tissue disorders) | 1 (1)
Ulcerative Colitis (Gastrointestinal disorders) | 1 (1)
Thromboembolism (Blood and lymphatic system disorders) | 1 (1)
Erosive Gastropathy (Gastrointestinal disorders) | 1 (1)
Gastric Angiodysplasia (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2)
Clostridium Difficile (Infections and infestations) | 1 (1)
Liver Failure (Hepatobiliary disorders) | 3 (3)
Jaundice (Hepatobiliary disorders) | 2 (2)
Heart Insufficiency (Cardiac disorders) | 1 (1)
Acute Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aplastic Bone Marrow (Blood and lymphatic system disorders) | 1 (1)
Gout Attack (Musculoskeletal and connective tissue disorders) | 1 (1)
Ankle Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hepatic Encephalopathy (Hepatobiliary disorders) | 5 (5)
Fatal Cardiac Arrest (Cardiac disorders) | 1 (1)
Fatal Ischemic Heart Disease (Cardiac disorders) | 1 (1)
Collapse (Nervous system disorders) | 1 (1)
Retinal Vein Thrombosis (Vascular disorders) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Syncope (Nervous system disorders) | 4 (5)
Rectal Ulcer (Gastrointestinal disorders) | 1 (1)
Liver Dysfunction (Hepatobiliary disorders) | 1 (1)
Coma (Nervous system disorders) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Pulmonary Thromboembolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis Pain (General disorders) | 1 (1)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Edema (Blood and lymphatic system disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pericarditis Constrictive (Cardiac disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Function Liver Abnormal (Hepatobiliary disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Duodenal Ulcer (Gastrointestinal disorders) | 4 (4)
Fatal Subdural Bleeding (Blood and lymphatic system disorders) | 1 (1)
Fatal Brain Edema (Blood and lymphatic system disorders) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Infections and infestations) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Hepatic Infarction (Hepatobiliary disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fecal Incontinence (Gastrointestinal disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Erythropoiesis (Blood and lymphatic system disorders) | 1 (1)
Hepatic Necrosis (Hepatobiliary disorders) | 1 (1)
Portal Vein Thrombosis (Vascular disorders) | 1 (1)
Liver Hemorrhage (Hepatobiliary disorders) | 1 (1)
CRP Increased (Hepatobiliary disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Altered State of Consciousness (Nervous system disorders) | 1 (1)
Periapical Abscess (Infections and infestations) | 1 (1)
Pneumatosis Intestinalis with Pneumoperitoneum (Skin and subcutaneous tissue disorders) | 1 (1)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 (1)
Femoral Artery Occlusion (Vascular disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Cavitation of Pulmonary Hilar Mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Enterovaginal Fistula (Reproductive system and breast disorders) | 1 (1)
Enterocutaneous Fistula (Gastrointestinal disorders) | 1 (1)
Stroke (Cardiac disorders) | 1 (1)
Central Retinal Vein Occlusion (Vascular disorders) | 1 (1)
Nephrotic Syndrome (Renal and urinary disorders) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Transient Ischaemic Attack (Cardiac disorders) | 1 (1)
Ulcerative Keratitis (Eye disorders) | 1 (1)
Necrosis of a Pleural Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchopleural Fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1)
Variceal Haemorrhage (Vascular disorders) | 1 (1)
Multi Organ Failure (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Cerebral Seizure (Nervous system disorders) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1)
Squamous Cell Cancer of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hearing Loss (Ear and labyrinth disorders) | 1 (1)
Induration (Skin and subcutaneous tissue disorders) | 1 (1)
Hydronephrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib 400 mg (N=105)
Allergic Reaction (Immune system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
ALT, SGPT (Metabolism and nutrition disorders) | 1
Amenorrhea (Reproductive system and breast disorders) | 1
Anorexia (Gastrointestinal disorders) | 5
AST, SGOT (Metabolism and nutrition disorders) | 1
Atrial Tachycardia (Cardiac disorders) | 1
Bilirubin (Metabolism and nutrition disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 8
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Elevated LDH (Metabolism and nutrition disorders) | 1
Erythema Multiform (Skin and subcutaneous tissue disorders) | 9
Fatigue (General disorders) | 9
Fever Unknown Origin (General disorders) | 1
Fever Without Neutropenia (General disorders) | 1
Flushing (Skin and subcutaneous tissue disorders) | 1
Gastrointestinal (Gastrointestinal disorders) | 2
Hand-Foot Syndrome (Musculoskeletal and connective tissue disorders) | 15
Hematuria (Renal and urinary disorders) | 1
Hemoglobin (Metabolism and nutrition disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Cardiac disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypotension (Cardiac disorders) | 1
Metabolic Laboratory (Metabolism and nutrition disorders) | 1
Mood Alteration (Nervous system disorders) | 2
Mucositis (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 5
Nausea Alone (Gastrointestinal disorders) | 1
Neutrophils (Blood and lymphatic system disorders) | 1
Ocular Surface Disease (Eye disorders) | 1
Pain (Chest Wall) (Cardiac disorders) | 1
Pain (Head/Headache) (Nervous system disorders) | 2
Pain (NOS) (General disorders) | 1
Pain (Oral Cavity) (General disorders) | 2
Petechiae (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Itching (Skin and subcutaneous tissue disorders) | 1
Sore Throat (General disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Syndromes (other) (General disorders) | 1
Taste Alteration (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes